CLINICAL TRIAL: NCT02592941
Title: An Open Label, Expanded Access Protocol Intended to Provide Treatment With MP-104 (Deflazacort) to U.S. Children, Adolescents, and/or Adults With Duchenne Muscular Dystrophy
Brief Title: Deflazacort Expanded Access Program for Children, Adolescents and Adults With Duchenne Muscular Dystrophy
Status: Approved for marketing | Type: Expanded Access
Sponsor: PTC Therapeutics (Industry)
Collaborators: Parexel (Industry); Dohmen Life Science Services (Other)
Responsible Party: Sponsor
Other Study IDs: MP-104-CL-037
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — deflazacort

INTERVENTIONS:
Drug: Deflazacort — Deflazacort, a glucocorticoid with anti-inflammatory and immunosuppressive effects, is used in treating a variety of diseases. Pharmacologically it is an inactive pro-drug which is metabolized immediately to the active metabolite, 21 desacetyl-DFZ. The elimination of this metabolite is primarily via the urine in humans. Its potency is approximately 70 to 90% of prednisone and 6 mg of deflazacort has approximately the same anti-inflammatory potency as 5 mg of prednisolone or prednisone.
  Other Names: DFZ

SUMMARY:
The expanded access program will provide access to treatment with deflazacort in children, adolescent, and adult patients with DMD in the U.S. who are ineligible, unable, or otherwise unwilling to enroll in a clinical study examining the efficacy of deflazacort while a new drug application is under preparation and review. Enrollment is open to all eligible patients.

DETAILED DESCRIPTION:
Deflazacort will be supplied free of charge and shipped directly to patients or caregivers, as appropriate. Treating physicians will continue to follow their standard of care activities and procedures for management of DMD. Treating physicians participating in the expanded access program are required to collect/document any patient or caregiver reported safety events and report to the sponsor..

ELIGIBILITY:
Main Inclusion Criteria:

* Confirmed diagnosis of Duchenne muscular dystrophy
* The patient is ≥ 5 years old
* Current on all childhood vaccinations including the chicken pox vaccine

Main Exclusion Criteria:

* History or current medication condition that could affect safety or poses an additional risk
* Hypersensitivity or allergic reaction to steroids or their formulations

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCLA Health, Los Angeles, California
  - Childrens Hospital of Orange County, Orange, California
  - UC Davis Medical Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Clinical Research Center, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Shriner's Hospital for Children - Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta- Scottish Rite, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Shriner's Hospital for Children - Chicago, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University- Children's Hospital of Michigan, Detroit, Michigan
  - Helen DeVos Children's Hospital Neurology Clinic, Grand Rapids, Michigan
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Las Vegas Clinic, Las Vegas, Nevada
  - Neurosciences Institute, Neurology-Charlotte, Charlotte, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Shriner's Hospital for Children, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Wesley Neurology Clinic, Cordova, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center - San Antonio, San Antonio, Texas
  - University of Virginia Children's Hospital, Charlottesville, Virginia
  - Children's Specialty Group, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- See also: www.accessdmd.com — http://www.accessdmd.com